CLINICAL TRIAL: NCT04943926
Title: Dietary Strategies for Remission of Type 2 Diabetes - a Randomized Controlled Trial (CARBCOUNT)
Brief Title: Dietary Strategies for Remission of Type 2 Diabetes
Acronym: CARBCOUNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Karolinska Institutet (Other); University of Glasgow (Other); University of Copenhagen (Other); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARBCOUNT Multicenter RCT
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity; Hypertension; Glucose Intolerance; Insulin Resistance; Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: Low-carbohydrate high-fat diet; Energy restricted diet; Lifestyle change; Ketogenic diet; Total meal replacement
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Hypertension; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomised controlled trail (RCT)
Who Masked: Outcomes Assessor
Masking Description: We will use an independent statistician who will analyse the data anonymously and be blinded to information regarding dietary arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy Restricted Diet (Active Comparator): A nutritional complete formula diet for 3 months followed by an energy restricted diet for 12 months.
  Interventions: Other: Energy restricted diet
- Continuous LCHF Diet (Experimental): A very low-carbohydrate high-fat ketogenic diet (VLCHF) diet for 3 months, followed by a low-carbohydrate high-fat diet (LCHF) for 12 months.
  Interventions: Other: Low carbohydrate high fat diet

INTERVENTIONS:
Other: Energy restricted diet — Nutritional complete formula diet followed by an energy restricted diet
  Arms: Energy Restricted Diet
Other: Low carbohydrate high fat diet — Very low-carbohydrate high-fat ketogenic diet (VLCHF) diet followed by a low-carbohydrate high-fat diet (LCHF)
  Arms: Continuous LCHF Diet

SUMMARY:
In this project, the investigators will perform a multicenter randomised controlled trial to determine whether advice to consume a moderate, whole food-based low-carbohydrate high-fat (LCHF) ad libitum diet (CarbCount program) can produce and maintain equal remission rates of type 2 diabetes (T2D) as a nutritionally complete very-low-calorie formula diet followed by a energy-restrictive (i.e., calorie counting) diet (DiRECT principles). Within the principles of each approach, the dietary goals and change will be adjusted according to individual needs/capabilities conducive to long-term adherence. Furthermore, the investigators aim to determine whether the rate of diet-induced remission is reflected in/can be predicted by baseline or diet-induced changes in glucose variability (e.g., time-in-range measured by continuous glucose monitoring) and other factors such as anthropometric changes and genetic susceptibility. Each center will also conduct locally-lead standalone mechanistic research, including analyses of intra-abdominal/hepatic fat accumulation, adipose tissue biopsies and/or measurements of energy metabolism. Additionally, changes in medication use, nutritional status, cardiovascular disease risk, as well as adverse events, will be monitored.

DETAILED DESCRIPTION:
At least 588 patients with T2D will be recruited, approximately 120-150 men and women at each research center. The participants will be randomised to 1) a nutritional complete formula diet for 3 months followed by an energy restricted diet for 12 months or 2) a very low-carbohydrate high-fat (VLCHF) diet for 3 months, followed by a low-carbohydrate high-fat diet (LCHF) for 12 months. Each of the diets will cover all basic requirements for essential nutrients including amino acids, fatty acids, vitamins and minerals. Participants will be encouraged to consume at least 200 g of vegetables per day. Furthermore, we will emphasize high-quality, minimally processed foods. In arm 2 they will receive advice to eat specific fat sources such as extra virgin olive oil, butter and high-fat cheeses.

The DiRECT trial showed remission in 46% of participants after 12 months. Assuming that both the DiRECT program and LCHF dietary strategies yield a 45% chance of T2D remission after 15 months, it is calculated (using nQuery v8) that each group needs 235 participants to complete the trial. This sample size yields 90% statistical power to conclude, with respect to the primary outcome, whether the CarbCount Program is no more than 15% more or less effective than the DiRECT principles (equivalence study, one-sided p-value at 0.025). To allow for expected loss to follow-up (estimated at 20%), each of the arms needs at least 294 participants for a total of 588.

Participants will have access to electronic platforms that include an online database of recipes (breakfast, easy-to-cook lunches, snacks, dinners, and food for special occasions). The platforms will facilitate planning of week menus, and include an e-learning course covering topics such as how to cook and prepare foods, meal planning, dining out, sleep and individual aspects that challenge habit change. If the participants are failing in their efforts to establish or maintain lifestyle change, they will be encouraged to seek possible solutions in the e-learning courses or to contact one of the study's health educators and/or dietitians. Specific rescue plans involving direct contact with study staff will be implemented if a participant regains more than 2 kg or experiences T2D relapse.

After individual assessment by a doctor, the participants will be taken off diabetes medication upon starting the diet, and be asked to self-monitor blood sugar changes during the first 2 weeks on the diet, followed by a consultation that includes evaluation of these changes. The need of reintroduction of medication will be done in consultation with the study doctor at least every 3 months.

Between visits, the participants will complete dietary assessments and an e-learning course, and at least once a month have follow-ups with dietitians/health educators and/or online group workshops.

The study will enroll eligible participants to the study continuously, until the total number of participants needed for the study is reached. Each participant will follow their own timeline, and attend visits at the study center at baseline, 3, 9 and 15 months.

During 2 weeks before each visit, participants will wear a continuous glucose monitor (CGM) and record food intake for at least 3 consecutive days during this period.

Measurements during visits will include anthropometric variables/body composition and energy expenditure, blood, saliva, urine and stool samples will be collected, and participants will be asked to fill out questionnaires on physical activity, sleep pattern, meal frequency, quality of life, problem areas in diabetes, eating efficacy and eating behaviors. They will also have a consultation with a registered dietitian and meet with the study medical doctor when needed.

A blinded statistician will perform the statistical analyses for the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥48 mmol/mol (with or without medical treatment)
* Less than 10 years since the diagnosis of T2D
* BMI ≥27 kg/m2 (≥25 kg/m2 for Asians)

Exclusion Criteria:

* Treatment with insulin >25 IU
* HbA1c concentration of 12% or more (≥108 mmol/mol)
* Insulin to C-peptide ratio <0.8 (indicative of insulin deficiency)
* Myocardial infarction within the previous 6 months, and severe or unstable heart failure or other severe diseases including cancer, psychiatric/eating disorders, severe depression and substance abuse

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes remission | 15 months
  Number of patients with diabetes remission, defined as no use of glucose-lowering drugs and HbA1c <48 mmol/mol (<6.5%) at 15 months

SECONDARY OUTCOMES:
Diabetes remission without anti-diabetes medications | 3, 9 and 15 months
  Number of patients with HbA1c <48 and <42 mmol/mol at 3, 9 and 15 months, both on and off anti-diabetes medication (metformin etc.)
Changes in HbA1c and fasting glucose concentrations from baseline | 3, 9 and 15 months
  HbA1c and fasting glucose concentrations (treatment targets in current clinical practice) measured in fasting blood samples
Changes in fasting insulin and insulin C-peptide concentrations from baseline | 3, 9 and 15 months
  Insulin and insulin C-peptide measured in fasting blood samples
Changes in estimated insulin resistance and beta cell function from baseline | 3, 9 and 15 months
  The HOMA2-calculator (https://www.dtu.ox.ac.uk/homacalculator/download.php) is used to estimate insulin resistance and beta cell function based on fasting glucose and C-peptide concentrations
Changes from baseline in the frequency of diabetes- and antihypertensive medication usage | 3, 9 and 15 months
  The number of diabetes- and antihypertensive medications used/reintroduced by each study visit counted and compared between groups
Changes in eating behaviour from baseline and throughout the study | 3, 9 and 15 months
  Eating behaviour measured by the The Weight Efficacy Lifestyle Questionnaire - Short form (WEL-SF). The questionnaire contains 8 items on a 10-point response scale (ranging from not at all confident/very confident). Responses to each item are given a score between 0-10, summed together and transformed to percentages. Changes in these scores will be compared between the study groups for the respective time-points throughout the intervention.
Changes in eating self-efficacy (Three-Factor Eating Questionnaire, TFEQ) | 3, 9 and 15 months
  Eating self-efficacy assessed by the Three-Factor Eating Questionnaire (TFEQ), which measures 3 aspects of eating behaviour: cognitive restraint, uncontrolled eating, and emotional eating. The questionnaire consists of 18 items on a 4-point response scale ( ranging from definitely true/mostly true/mostly false/definitely false). Responses to each item are given a score between 1 and 4 and and total scores are summed by the 3 measured aspects mentioned above. The raw scale scores are transformed to a 0-100 scale. Changes in these scores will be compared between the study groups for the respective time-points throughout the intervention.
Changes in quality of life | 3, 9 and 15 months
  Quality of life measured by the EQ-5D-5L questionnaire, which includes 5 dimensions: mobility, self-care, usual activities, pain /discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The levels are scored with a 1-digit number and the digits for the five dimensions are combined into a 5-digit number that describes the patient's health state. We will compare change at all timepoints between groups using both the 1-digit and the 5-digit number.
  The questionnaire includes the patient's self-rated health on a Visual analog scale (VAS) ranging from 0-100. The endpoints are labelled "The best health you can imagine" and "The worst health you can imagine". The scale will be transposed into percentages and the percent change will be compared between the study groups.

OTHER OUTCOMES:
Rates of T2D remission dependent on polygenic risk scores for T2D | 3, 9 and 15 months
  Polygenic risk scores are calculated based on the latest GWAS data for T2D, and rates of remission compared between patients with the top 20% high- and top 20% low scores, for all participants combined and the respective diets separately
Changes in ectopic fat accumulation from baseline | 3, 9 and 15 months
  Body fat measured by MRI (abdominal adipose tissue distribution, hepatic-, intramuscular-, pericardial- and pancreatic fat)
Changes in liver fibrosis and steatosis from baseline | 3, 9 and 15 months
  Liver fibrosis and steatosis measured by ultrasound-based transient elastography
Changes in markers of liver function from baseline | 3, 9 and 15 months
  Alanine transaminase (ALT), C-reactive protein (CRP) and other markers of liver function measured in fasting blood samples
Changes in inflammatory markers from baseline | 3, 9 and 15 months
  Circulating concentrations of selected markers of inflammation measured in fasting blood samples by ELISA
Changes in blood pressure and pulse from baseline | 3, 9 and 15 months
  Blood pressure and pulse measured after 10 minutes in resting position
Change in CVD risk (NORRISK) from baseline | 3, 9 and 15 months
  NORRISK calculated by the most current NORRISK calculator (https://hjerterisiko.helsedirektoratet.no/)
Changes in total-, low-density lipoprotein (LDL), high-density lipoprotein (HDL) and very-low-density (VLDL) cholesterol concentrations from baseline | 3, 9 and 15 months
  Blood lipids measured in fasting blood samples
Changes in triacylglycerols (TGs) and TG/HDL-C ratio from baseline | 3, 9 and 15 months
  Blood lipids measured in fasting blood samples
Changes in lipoprotein subfractions from baseline | 3, 9 and 15 months
  Lipoprotein particle numbers and sizes (small/medium/large LDL, IDL, HDL, VLDL) measured in fasting blood samples
Changes in apolipoproteins from baseline | 3, 9 and 15 months
  Apolipoproteins (including apoB, apoAs, ApoCs) measured in fasting blood samples
Changes in micronutrient status from baseline | 3, 9 and 15 months
  Micronutrients measured in the circulation in fasting blood samples
Changes in gut and oral microbiota from baseline | 3, 9 and 15 months
  Gut and oral microbiota measured by 16S sequencing in feces and saliva, respectively
Changes in appetite/satiety and ketones from baseline | 3, 9 and 15 months
  Ghrelin and ketones measured in fasting blood samples, and correlations in the change of ghrelin and ketones (beta-hydroxybutyrate and acetoacetate) from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Science, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No